CLINICAL TRIAL: NCT04880473
Title: A Minimal-Risk, Multi-Center, Prospective, Clinical Trial to Evaluate the PrevisEA Device for Predicting Gastrointestinal Impairment
Brief Title: Evaluation of the PrevisEA Device for Predicting Gastrointestinal Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Entac Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Entac-PrevisEA-001
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Complication
Keywords: Postoperative ileus; Postoperative bowel obstruction; Emesis; Reversal of diet; Nasogastric tube; Abdominal sounds; Gastrointestinal impairment; Elective intestinal resection
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrevisEA device (Experimental): The PrevisEA device is placed and activated on the patient's abdomen immediately post-op (within 1 hour of the completion of surgery) and maintained in position for at least 12 hours, counting the number of times MH4 is detected within a four-minute period at hourly intervals. The device determines the MH4 biomarker counts at each hourly collection point and the data are stored on the device. For this clinical trial, the display is obscured. Therefore, no value will be displayed for interpretation since this is a non-intervention trial and the device is not intended to affect or influence the standard of care for study participants.
  Interventions: Device: PrevisEA device

INTERVENTIONS:
Device: PrevisEA device — The PrevisEA device is placed and activated on the patient's abdomen immediately post-op (within 1 hour of the completion of surgery) and maintained in position for at least 12 hours, counting the number of times MH4 is detected within a four-minute period at hourly intervals. The device determines the MH4 biomarker counts at each hourly collection point and the data are stored on the device. Under normal conditions, transformations of the data are visualized on the display. For this clinical trial, the display is obscured. Therefore, no value will be displayed for interpretation since this is a non-intervention trial and the device is not intended to affect or influence the standard of care for study participants.

SUMMARY:
PrevisEA is a noninvasive, disposable device that uses audio spectral analysis of sounds produced by the gastrointestinal tract to predict gastrointestinal impairment (GII). GII is most commonly associated with postoperative ileus (POI), but could be the result of other causes, such as early postoperative bowel obstruction. GII is defined as failure of successful early oral re-feeding in a subject undergoing major abdominal surgery. For subjects who are allowed to resume a diet during the first 24 hours after surgery, a failure to successfully orally re-feed a subject is defined as presentation with emesis, requiring a reversal of diet, or the placement of a nasogastric tube on first postoperative day or later.

The device is considered non-significant risk (NSR). The device does not inform medical decisions in this study. Researchers will be blinded to results of the device during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 90 years
2. Patient undergoing elective intestinal resection surgery including open, laparoscopic, robotic, or hand-assist technique for:

   1. Segmental ileocolic resection with or without diversion
   2. Segmental colon resection with or without diversion
   3. Segmental coloproctectomy with or without diversion
   4. Low anterior resection with or without diversion
   5. Abdominoperineal resection
   6. Total abdominal colectomy with or without diversion
   7. Proctocolectomy with or without end ileostomy or diversion
   8. Closure of end colostomy (Hartmann's reversal)

Exclusion Criteria:

1. Allergies to any of the device components (i.e., adhesive)
2. Inability to have prototype device applied to their abdominal wall due to disease conditions or surgical alterations(e.g., fistulas, stomas, drains, etc.)
3. Patients undergoing:

   1. Small bowel resection without colonic resection
   2. Transanal proctectomy without transabdominal approach
   3. Perineal proctosigmoidectomy
   4. Closure of loop colostomy or ileostomy
4. Patients with preoperative evidence of an anastomotic leak, deep wound infection, organ space infection, or urinary tract infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the PrevisEA device | 1-14 days
  The performance (accuracy) of the device in predicting development of GII will be assessed through evaluation of the primary outcome measures of sensitivity and specificity for the device.

SECONDARY OUTCOMES:
Positive predictive value (PPV) | 1-14 days
  Measures will be analyzed by using available data only
Negative predictive value (NPV) | 1-14 days
  Measures will be analyzed by using available data only
Overall percent agreement (OPA) | 1-14 days
  Measures will be analyzed by using available data only

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Adventist Health System/Sunbelt, Inc. d/b/a AdventHealth Orlando, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Spectrum Health Blodgett Hospital, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No